CLINICAL TRIAL: NCT02353299
Title: Phase IV 4 Way Crossover Study to Assess and Compare the Effect of a Single Nighttime Administration of Zolpidem, Silenor and Placebo on Arousability, Ataxia/Balance and Cognitive Performance in Healthy Volunteers.
Brief Title: Assess the Effect of Zolpidem, Silenor & Placebo on Arousability, Ataxia/Balance & Cognition in Healthy Volunteers
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Currax Pharmaceuticals (Industry)
Collaborators: Henry Ford Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Diagnostic
Other Study IDs: PT-D1402
Record Dates: First submitted 2015-01-23; First posted 2015-02-02 (Estimated); Results first posted 2017-12-07 (Actual); Last update posted 2018-01-02 (Actual); Status verified 2017-12

CONDITIONS: Healthy
Keywords: Cognition; Balance
MeSH Terms: interventions — Doxepin; Zolpidem

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Silenor 6 mg (DXP-4H) (Active Comparator): Silenor 6 mg single nightime dose- 4 hour post dose arousability and cognitive assessments
  Interventions: Drug: Silenor 6 mg; Drug: zolpidem 10 mg; Drug: Placebo
- Placebo (PBO-4H) (Placebo Comparator): placebo single nightime dose -4 hour post dose arousability and cognitive assessments
  Interventions: Drug: Silenor 6 mg; Drug: zolpidem 10 mg; Drug: Placebo
- Zolpidem 10 mg (ZOL-1.5H) (Active Comparator): zolpidem 10 mg single nightime dose - 1.5 hour arousability and cognitive assessments
  Interventions: Drug: Silenor 6 mg; Drug: zolpidem 10 mg; Drug: Placebo
- Placebo (PBO-1.5H) (Placebo Comparator): placebo single nightime dose -1.5 hour arousability and cognitive assessments
  Interventions: Drug: Silenor 6 mg; Drug: zolpidem 10 mg; Drug: Placebo

INTERVENTIONS:
Drug: Silenor 6 mg — Silenor 6 mg single nighttime dose.
  Other Names: doxepin
Drug: zolpidem 10 mg — Zolpidem 10 mg single nighttime dose
  Other Names: zolpidem
Drug: Placebo — placebo single nighttime dose-1.5 hours
Drug: Placebo — placebo single nighttime dose-4 hours

SUMMARY:
This is a Phase IV, randomized, double-blind, placebo-controlled, four-arm crossover study. The study will assess the effects of a single dose of Silenor 6 mg compared with matching placebo and a single dose of zolpidem 10 mg compared to its matching placebo at the respective T-max in normal healthy adult male volunteers. The study will be conducted in approximately 52 male subjects

DETAILED DESCRIPTION:
Subjects will be screened and asked to complete sleep disorders questionnaires and a sleep diary to establish normal sleep patterns and to rule out any sleep disorder.

Eligible subjects will be scheduled for a Screening PSG to rule out PLMS, sleep apnea and other sleep disorders.

Subjects who meet the screening PSG criteria will be randomly assigned to a treatment sequence order that involves both the study drug and the time subjects are awakened in the middle-of-the-night using a crossover study design. These four sequences include Silenor 6 mg with a middle-of-the-night awakening at 4 hours (DXP-4H), zolpidem 10 mg with a middle-of-the-night awakening at 1.5 hours (ZOL-1.5H), placebo with a middle-of-the-night awakening at 4 hours (PBO-4H), and placebo with a middle-of-the-night awakening at 1.5 hours (PBO-1.5H). Study drug will be administered under fasted conditions (at least 4 hours) as a single dose at bedtime (approximately 2300 hours), and each subject will receive one dose of each active drug (Silenor 6 mg and zolpidem 10 mg), and two doses of placebo during the treatment period.

Safety assessments will be performed throughout the study.

During the night of assessment, subjects will be awoken at the estimated T-max of the active drugs, with a matching placebo group awakened at each of these time points with the same arousability protocol. Arousability will be assessed using the Auditory Awakening Threshold test (AAT) .

Once the Auditory Awakening Threshold has been determined, subjects will perform a Tandem Walk assessment followed by the Berg Balance Scale (BBS) and finally by Free Recall Memory testing.

Subjects will be discharged from the sleep center once all assessments have been completed. A final study visit will be performed for subjects either after they have completed all four Treatment Periods or they have prematurely discontinued the study.

ELIGIBILITY:
Inclusion Criteria:

* Be in good general health as determined by the investigator;
* Have a 3-month history of a normal nightly sleep pattern based on the subject's self report ;
* A usual time in bed
* A regular bedtime between 2200 and 2400 hours
* No habitual daytime napping;
* Epworth Sleepiness Scale score ≤ 10;
* Be able to read, understand, and provide written/dated informed consent before enrolling in the study, and must be willing and able to comply with all study procedures;
* Be able to follow verbal and written instructions provided in English

Exclusion Criteria:

* Have a body mass index (BMI) >35 kg/m2
* Have symptoms consistent with the diagnosis of any sleep disorder (e.g., insomnia, sleep apnea, narcolepsy, periodic leg movements, or restless leg syndrome);
* On screening PSG AHI > 10 or PLMAI >10;
* Have a known or suspected diagnosis of Acquired Immune Deficiency Syndrome (AIDS), or have tested seropositive for human immunodeficiency virus (HIV) antibody or antigen previously;
* Have any clinically significant abnormal finding in physical examination, neurological assessment, vital signs, elevated body temperature, or clinical laboratory tests, as determined by the Investigator;
* Have a known exaggerated pharmacological sensitivity, hypersensitivity, or history of a clinically significant adverse reaction to zolpidem;
* Have a known or exaggerated pharmacological sensitivity, hypersensitivity, or intolerance to doxepin HCl, any tricyclic antidepressant, or antihistamine;
* Currently taking cimetidine or a monoamine oxidase inhibitor (MAOI);
* Current diagnosis of severe urinary retention;
* Current diagnosis of untreated glaucoma;
* Intends to use any medication including over-the-counter (OTC) medications that would interfere with normal sleep architecture (such as systemic steroids, beta-adrenergic blockers, amphetamines, modafinil, etc.);
* Self-reports use of products containing nicotine of greater than 15 cigarettes daily, or cannot avoid products containing nicotine during the normal sleep periods;
* Self report consumption of more than five alcoholic beverages on any one day or greater than 14 alcoholic beverages weekly over the past week;
* Have a history of epilepsy or serious head injury;
* Used CYP450 2D6 inducers or inhibitors within 7 days before screening;
* Have used prescribed or OTC medications within 30 days of screening (Day 0) or intend to use any prescription or OTC medication during the study that may interfere with the evaluation of the study drug.
* Have used an investigational drug within 30 days or five half lives (whichever is longer) before screening, or plans to use an investigational drug during the study or have used doxepin or zolpidem previously.
* Score of < 40 on the BBS at screening

Ages: 21 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 52 (Actual)
Dates: Start 2015-01; Primary Completion 2016-01 (Actual); Study Completion 2016-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chris Drake, PhD, Principal Investigator — Henry Ford Hospital Sleep Disorder Research Center
Locations (1):
- Henry Ford Hospital Sleep Disorders & Research Center, Novi, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Davis KL, Charey D, Cuyle JT, Nemeroff C. Neuropsychopharmacology, The Fifth Generation of Progress. 2002; Section 13: 1938-1939
- [Background] Silenor [prescribing information]. Pernix Pharmaceuticals, Inc., San Diego, CA; March 2010.
- [Background] Sanofi-Synthelabo. Ambien (zolpidem tartrate) complete prescribing information. 2002.
- [Background] Johns MW. A new method for measuring daytime sleepiness: the Epworth sleepiness scale. Sleep. 1991 Dec;14(6):540-5. doi: 10.1093/sleep/14.6.540. PMID 1798888
- [Result] Rechtschaffen A, Kales A, eds. A Manual of Standardized Terminology, Techniques and Scoring System for Sleep Stages of Human Subjects. Los Angeles, Calif; Brain Information Service/Brain Research Institute, UCLA; 1968
- [Result] Berg Balance Scale (BBS)
- [Result] Mintzer MZ, Griffiths RR. Selective effects of zolpidem on human memory functions. J Psychopharmacol. 1999;13(1):18-31. doi: 10.1177/026988119901300103. PMID 10221356
- [Result] Gottlieb DJ, Yenokyan G, Newman AB, O'Connor GT, Punjabi NM, Quan SF, Redline S, Resnick HE, Tong EK, Diener-West M, Shahar E. Prospective study of obstructive sleep apnea and incident coronary heart disease and heart failure: the sleep heart health study. Circulation. 2010 Jul 27;122(4):352-60. doi: 10.1161/CIRCULATIONAHA.109.901801. Epub 2010 Jul 12. PMID 20625114
- [Result] Chung F, Yegneswaran B, Liao P, Chung SA, Vairavanathan S, Islam S, Khajehdehi A, Shapiro CM. STOP questionnaire: a tool to screen patients for obstructive sleep apnea. Anesthesiology. 2008 May;108(5):812-21. doi: 10.1097/ALN.0b013e31816d83e4. PMID 18431116
- [Derived] Drake CL, Durrence H, Cheng P, Roth T, Pillai V, Peterson EL, Singh M, Tran KM. Arousability and Fall Risk During Forced Awakenings From Nocturnal Sleep Among Healthy Males Following Administration of Zolpidem 10 mg and Doxepin 6 mg: A Randomized, Placebo-Controlled, Four-Way Crossover Trial. Sleep. 2017 Jul 1;40(7). doi: 10.1093/sleep/zsx086. PMID 28575467

RESULTS

PARTICIPANT FLOW:
Groups:
- PBO-4H Then PBO-1.5H Then DXP-4H Then ZOL-1.5H: Period 1: Doxepin-matching placebo-single nighttime dose Period 2: Zolpidem-matching placebo-single nighttime dose Period 3: Doxepin 6mg-single nighttime dose Period 4: Zolpidem 10 mg-single nighttime dose
- PBO-1.5H Then ZOL-1.5H Then PBO-4H Then DXP-4H: Period 1: Zolpidem-matching placebo-single nighttime dose Period 2: Zolpidem 10 mg-single nighttime dose Period 3: Doxepin-matching placebo-single nighttime dose Period 4: Doxepin 6mg-single nighttime dose
- ZOL-1.5H Then DXP-4H Then PBO-1.5H Then PBO-4H: Period 1: Zolpidem 10mg-single nighttime dose Period 2: Doxepin 6mg-single nighttime dose Period 3: Zolpidem-matching placebo-single nighttime dose Period 4: Doxepin-matching placebo-single nighttime dose
- DXP-4H Then PBO-4H Then ZOL-1.5H Then PBO-1.5H: Period 1: Doxepin 6mg-single nighttime dose Period 2: Doxepin-matching placebo-single nighttime dose Period 3: Zolpidem 10mg-single nighttime dose Period 4: Zolpidem-matching placebo-single nighttime dose
Period: First Intervention (1 Night)
Arm/Group | PBO-4H Then PBO-1.5H Then DXP-4H Then ZOL-1.5H | PBO-1.5H Then ZOL-1.5H Then PBO-4H Then DXP-4H | ZOL-1.5H Then DXP-4H Then PBO-1.5H Then PBO-4H | DXP-4H Then PBO-4H Then ZOL-1.5H Then PBO-1.5H
Started | 13 | 13 | 13 | 13
Completed | 13 | 13 | 13 | 13
Not Completed | 0 | 0 | 0 | 0
Period: Second Intervention (1 Night)
Arm/Group | PBO-4H Then PBO-1.5H Then DXP-4H Then ZOL-1.5H | PBO-1.5H Then ZOL-1.5H Then PBO-4H Then DXP-4H | ZOL-1.5H Then DXP-4H Then PBO-1.5H Then PBO-4H | DXP-4H Then PBO-4H Then ZOL-1.5H Then PBO-1.5H
Started | 13 | 13 | 13 | 13
Completed | 13 | 13 | 13 | 13
Not Completed | 0 | 0 | 0 | 0
Period: Third Intervention (1 Night)
Arm/Group | PBO-4H Then PBO-1.5H Then DXP-4H Then ZOL-1.5H | PBO-1.5H Then ZOL-1.5H Then PBO-4H Then DXP-4H | ZOL-1.5H Then DXP-4H Then PBO-1.5H Then PBO-4H | DXP-4H Then PBO-4H Then ZOL-1.5H Then PBO-1.5H
Started | 13 | 13 | 13 | 13
Completed | 13 | 13 | 13 | 13
Not Completed | 0 | 0 | 0 | 0
Period: Fourth Intervention (1 Night)
Arm/Group | PBO-4H Then PBO-1.5H Then DXP-4H Then ZOL-1.5H | PBO-1.5H Then ZOL-1.5H Then PBO-4H Then DXP-4H | ZOL-1.5H Then DXP-4H Then PBO-1.5H Then PBO-4H | DXP-4H Then PBO-4H Then ZOL-1.5H Then PBO-1.5H
Started | 13 | 12 (One patient withdrawn from study prior to start of fourth intervention.) | 13 | 13
Completed | 13 | 12 | 13 | 13
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Subjects were healthy males
Groups:
- All Study Participants: A single group of subjects were recruited and assigned all study treatments in random order
Arm/Group | All Study Participants
Number analyzed (Participants) | 52
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 52
  >=65 years | 0
Sex/Gender, Customized [Count of Participants; unit: Participants]
  male | 52
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 5
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 30
  More than one race | 0
  Unknown or Not Reported | 14
Region of Enrollment [Number; unit: participants]
  United States | 52

OUTCOME MEASURES:

1. Primary Outcome: Auditory Arousal Threshold (AAT) at T-max
Description: AAT will performed at T-max for Silenor and matching placebo at 4 hours post dose. Assessments performed at t max for zolpidem and placebo at 1.5 hours post dose.
  An acoustic stimulus (1000 Hz tone) was presented through audiometric earphones (E-A-RTone 3A Insert Earphones). Tones began at 30 dB and increased by 5 dB until the participant woke up or the maximum dB-level (110 dB) was reached.
Time Frame: at either 1.5 or 4 hours post dose
Measure: Mean (Standard Deviation); unit: Decibels (dB)
Arm/Group | Silenor 6 mg (DXP-4H) | Placebo (PBO-4H) | Zolpidem 10 mg (ZOL-1.5H) | Placebo (PBO-1.5H)
Number analyzed (Participants) | 51 | 52 | 52 | 52
Decibels (dB) | 85.2 (11.8) | 78.0 (18.6) | 103.2 (11.8) | 84.7 (17.1)

2. Secondary Outcome: Tandem Walk Step-Offs
Description: Tandem walk will be performed at T-max for Silenor and matching placebo at 4 hours post dose and at 1.5 hours post dose for zolpidem 10 mg and matching placebo.
  Fall risk as impacted by balance was measured using the Tandem Walk Test (TWT), which assesses balance via a method of walking in which the toes of the back foot must touch the heel of the front foot at each step; this elicits postural control by reducing the base of support compared to normal walking. Endpoints were the number of step-offs from the beam.
Time Frame: at either 1.5 or 4 hours post dose
Measure: Mean (Standard Deviation); unit: number of step offs
Arm/Group | Placebo (PBO-4H) | Silenor 6 mg (DXP-4H) | Zolpidem 10 mg (ZOL-1.5H) | Placebo (PBO-1.5H)
Number analyzed (Participants) | 52 | 51 | 52 | 52
number of step offs | 0.9 (1.4) | 1.5 (2.4) | 8.1 (8.0) | 1.0 (1.3)

3. Secondary Outcome: Tandem Walk Duration Over Five Trials
Description: Tandem walk will be performed at T-max for Silenor and matching placebo at 4 hours post dose and at 1.5 hours post dose for zolpidem 10 mg and matching placebo.
  Fall risk as impacted by balance was measured using the Tandem Walk Test (TWT), which assesses balance via a method of walking in which the toes of the back foot must touch the heel of the front foot at each step; this elicits postural control by reducing the base of support compared to normal walking. Endpoint: mean completion duration over five trials.
Time Frame: at either 1.5 or 4 hours post dose
Measure: Mean (Standard Deviation); unit: Seconds
Arm/Group | Placebo (PBO-4H) | Silenor 6 mg (DXP-4H) | Zolpidem 10 mg (ZOL-1.5H) | Placebo (PBO-1.5H)
Number analyzed (Participants) | 52 | 51 | 52 | 52
Seconds | 4.82 (1.68) | 4.97 (1.57) | 6.69 (2.60) | 4.83 (1.60)

4. Secondary Outcome: Berg Balance Test
Description: Berg Balance will be performed at T-max for silenor and matching placebo at 4 hours post dose and at 1.5 hours post dose for zolpidem 10 mg and matching placebo.
  Fall risk as impacted by gait was measured using the Berg Balance Scale (BBS). The BBS is a widely used clinical test of static and dynamic balance abilities. Comprising of 14 simple balance-related tasks, ranging from standing up from a sitting position to standing on one foot, the BBS takes 15-20 minutes to complete. Each component task is scored on a Likert scale: 0 (unable to perform) to 4 (performed independently). The sum of component scores yields the final BBS score (0-20: high fall risk; 21-40: medium fall risk; 41-56: low fall risk).
Time Frame: at either 1.5 or 4 hours post dose
Measure: Mean (Standard Deviation); unit: sum of component scores
Arm/Group | Silenor 6 mg (DXP-4H) | Placebo (PBO-4H) | Zolpidem 10 mg (ZOL-1.5H) | Placebo (PBO-1.5H)
Number analyzed (Participants) | 51 | 52 | 52 | 52
sum of component scores | 54.5 (1.9) | 55.1 (1.4) | 51.4 (4.3) | 55.1 (1.4)

5. Secondary Outcome: Immediate Free Recall Task
Description: Immediate Free Recall will be performed at T-max for silenor and matching placebo at 4 hours post dose and at 1.5 hours post dose for zolpidem 10 mg and matching placebo.
  Free Recall is a basic paradigm in the psychological study of memory. In this paradigm, participants were presented with a total of 16 words serially. They were informed prior to the task that memory for the presented words would be tested later in the session.
Time Frame: directly after the encoding task
Measure: Mean (Standard Deviation); unit: Number of words
Arm/Group | Silenor 6 mg (DXP-4H) | Placebo (PBO-4H) | Zolpidem 10 mg (ZOL-1.5H) | Placebo (PBO-1.5H)
Number analyzed (Participants) | 51 | 52 | 52 | 52
Number of words | 7.86 (3.20) | 8.14 (2.99) | 4.78 (3.42) | 7.71 (3.12)

6. Secondary Outcome: Delayed Free Recall Task
Description: Delayed Free Recall Task was performed 15 minutes after final awakening the morning
  Free Recall is a basic paradigm in the psychological study of memory. In this paradigm, participants were presented with a total of 16 words serially. They were informed prior to the task that memory for the presented words would be tested later in the session. Participants were asked to recall as many words as they can 15 minutes after final awakening in the morning
Time Frame: 15 minutes after final awakening the morning
Measure: Mean (Standard Deviation); unit: Number of words
Arm/Group | Silenor 6 mg (DXP-4H) | Placebo (PBO-4H) | Zolpidem 10 mg (ZOL-1.5H) | Placebo (PBO-1.5H)
Number analyzed (Participants) | 51 | 52 | 52 | 52
Number of words | 6.78 (3.68) | 7.02 (3.59) | 2.24 (2.77) | 6.51 (3.48)

7. Secondary Outcome: Number of Participants With Adverse Events
Description: Adverse events were defined by any negative event experienced by a participant during the study (assessed in the morning prior to participants leaving the lab) and included the washout period following each treatment.
Time Frame: throughout the study until the final study visit, up to 6 weeks
Measure: Number; unit: Participants
Arm/Group | Silenor 6 mg (DXP-4H) | Placebo (PBO-4H) | Zolpidem 10 mg (ZOL-1.5H) | Placebo (PBO-1.5H)
Number analyzed (Participants) | 51 | 52 | 52 | 52
Participants | 13 | 11 | 12 | 10

ADVERSE EVENTS:
Time Frame: Throughout the study period until the final study visit, up to 6 weeks.
Arm/Group | Silenor 6 mg (DXP-4H) | Placebo (PBO-4H) | Zolpidem 10 mg (ZOL-1.5H) | Placebo (PBO-1.5H)
All-Cause Mortality (participants affected / at risk) | 0/51 | 0/52 | 0/52 | 0/52
Serious Adverse Events (participants affected / at risk) | 0/51 | 0/52 | 0/52 | 0/52
Other Adverse Events (participants affected / at risk) | 13/51 | 11/52 | 12/52 | 10/52
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Silenor 6 mg (DXP-4H) (N=51) | Placebo (PBO-4H) (N=52) | Zolpidem 10 mg (ZOL-1.5H) (N=52) | Placebo (PBO-1.5H) (N=52)
Memory Impairment (Nervous system disorders) | 0 (0) | 1 (1) | 3 (3) | 0 (0)
Somnolence (Nervous system disorders) | 4 (4) | 4 (4) | 4 (4) | 0 (0)
Insomnia (Nervous system disorders) | 3 (3) | 3 (3) | 2 (2) | 2 (2)
Syncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Presyncope (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Fatigue/lethargy (General disorders) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Xerostomia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rigors (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Other (General disorders) | 2 (2) | 1 (1) | 1 (1) | 7 (7)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No